CLINICAL TRIAL: NCT06081244
Title: NeoAdjuvant Dynamic Marker - Adjusted Personalized Therapy Comparing Sacituzumab Govitecan Versus Sacituzumab Govitecan+Pembrolizumab in Low-risk, Triple-negative Early Breast Cancer (ADAPT-TN-III)
Brief Title: NeoAdj. Therapy Comparing Sacituzumab Govitecan (SG) vs. SG+Pembrolizumab in Low-risk, Triple-neg. EBC (ADAPT-TN-III)
Acronym: ADAPT-TN-III
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM13 (ADAPT-TN-III)
Record Dates: First submitted 2023-07-26; First posted 2023-10-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Triple Negative Breast Cancer
Keywords: TNBC; Early breast cancer; Sacituzumab govitecan; pembrolizumab; chemotherapy; low recurrence risk
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — sacituzumab govitecan; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a multicentre, interventional, prospective, two-arm, randomised, open-label, neoadjuvant, phase-II-trial evaluating the efficacy and safety of SG alone vs. SG+PEM in low-risk early TNBC in pre- and postmenopausal women.
Masking Description: Open Label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant treatment: 12 weeks (4 cycles) SG i.v. (Experimental): * Cohort 1a: In case of (near) cCR: end of treatment, followed by surgery
  * Cohort 1b: In case of cPR after 12 weeks: further 6 weeks (2 cycles) SG i.v., followed by surgery (use of core biopsy is allowed per investigator´s decision, if further NACT is planned) pCR dependent post-neoadjuvant treatment
  * In case of pCR: no further systemic treatment
  * In case of non-pCR: chemotherapy according to investigators decision, e.g., AC/EC q3w x 4, PAC/Carbo q1w x 12
  Interventions: Drug: Sacituzumab govitecan
- Neoadjuvant treatment: 12 weeks (4 cycles) SG+PEM i.v. (Experimental): * Cohort 2a: In case of (near) cCR: end of treatment, followed by surgery
  * Cohort 2b: In case of cPR after 12 weeks: 6 weeks (2 cycles) SG+PEM i.v., followed by surgery (use of core biopsy is allowed per investigator´s decision, if further NACT is planned) pCR dependent post-neoadjuvant treatment
  * In case of pCR: no further systemic treatment
  * In case of non-pCR: chemotherapy according to investigators decision, e.g., AC/EC q3w x 4, PAC/Carbo q1w x 12
  Interventions: Drug: Sacituzumab govitecan; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sacituzumab govitecan — 10 mg/kg twice on Days 1 and 8 of a continuous 21-day treatment cycle
  Other Names: Trodelvy
Drug: Pembrolizumab — 200 mg every 3 weeks (q3w)
  Other Names: Keytruda
  Arms: Neoadjuvant treatment: 12 weeks (4 cycles) SG+PEM i.v.

SUMMARY:
TNBC is known for poor prognosis, aggressive patterns of disease, and significant molecular heterogeneity. (Neo)adjuvant chemotherapy (NACT) is standard of care in all node-positive and in node-negative patients with a tumour size >5 mm according to current National Comprehensive Cancer Network (NCCN) guidelines. However, TNBC patients with lower stage disease do clearly have a better prognosis compared to more advanced stages. Patients with stage I-II node-negative disease have 3-5 year iDFS rates of 80-90% (with majority of relapses within the first three years) as shown in several trials.Although survival results appear much better in the lower vs. higher stages, there is a high clinical need in this most common group of TNBC patients in Western Europe and USA.

DETAILED DESCRIPTION:
About 15% of breast cancers lack both, expression of ER and PR receptors, and amplification/over-expression of HER2 receptors, and are thus described as triple negative breast cancer (TNBC). TNBC is known for poor prognosis, aggressive patterns of disease, and significant molecular heterogeneity. (Neo)adjuvant chemotherapy (NACT) is standard of care in all node-positive and in node-negative patients with a tumour size >5 mm according to current National Comprehensive Cancer Network (NCCN) guidelines. However, TNBC patients with lower stage disease do clearly have a better prognosis compared to more advanced stages. Patients with stage I-II node-negative disease have 3-5 year iDFS rates of 80-90% (with majority of relapses within the first three years) as shown in several trials. Our own results from the PlanB- and ADAPT-trials, and pooled analysis with SUCCESS C-trials show 3-year iDFS of 86-90% in node-negative TNBC with a tumour size < 3 cm. Although survival results appear much better in the lower vs. higher stages, there is a high clinical need in this most common group of TNBC patients in Western Europe and USA.

In the neoadjuvant setting, it has been shown that the prognosis of patients with TNBC is strongly dependent on their response to NACT: Patients achieving pathological complete response (pCR), or a near pCR (an excellent response after NACT (residual cancer burden (RCB) score 0-1), in some studies do have an excellent prognosis that is not significantly different from that observed in other breast cancer subtypes. However, patients with a less responsive disease (i.e., with RCB Score 2-3) suffer from a significantly worse prognosis compared to non-TNBC.

Chemotherapy in TNBC The optimal chemotherapy regimen for patients with TNBC remains to be identified. Standard anthracycline-taxane (A/T)-based NACT combinations render pCR rates between 25-50%. However, the survival impact of anthracyclines remains controversial due to conflicting results of different randomized trials. Adding carboplatin (carbo) to A/T-containing poly-NACT or use of dose-intensified poly-NACT significantly increases pCR-rates up to 49-60% in mostly stage II-III disease with conflicting survival results and higher toxicity. Hence, use of pragmatic taxane-carboplatin anthracycline-free combinations appears as an effective treatment option in TNBC instead of further treatment escalation. This probably is independent of the germline BRCA (gBRCA) status, due to its general chemo-predictive effect. Unfortunately, no prospective phase-III-data are available so far. However, indirect comparison between trials renders similar pCR rates in taxane-carboplatin based vs. A/T+/-carbo-based regimens in early TNBC.

In the ADAPT-TN neoadjuvant trial, the taxane-carbo arm (12-week nab-paclitaxel (nab-pac)+carbo) was well tolerable (only 10% SAE-rate), highly effective (pCR, ypT0/is/ypN0, of 46%) and superior to the gemcitabine (gem)-arm (nab-pac+gem, pCR of 29%). In this study, omission of further chemotherapy was allowed in patients with pCR after 12 weeks of therapy and was not associated with decreased survival after 3 years [5] and longer follow up.

Although a standard chemotherapy as well as optimal therapy duration are still to be defined, several studies are showing a comparable efficacy for longer vs. shorter adjuvant treatments in TNBC [3], as well as a similar efficacy regarding pCR in HR-negative (in contrast to HR-positive) early breast cancer (eBC) [26]. Moreover 6 vs. 4 cycles of the same chemotherapy (AC or pac weekly) yielded a similar survival outcome in eBC despite of HR-status. No such comparison regarding treatment duration is available for modern antibody-drug conjugates like sacituzumab govitecan (SG).

Therefore, an examination of shorter (12 weeks vs. 18 weeks) regimen as neoadjuvant treatment appears to be a very promising strategy at least in patients with lower risk disease or in elderly patients, who do not qualify for polychemotherapy treatments.

In the Keynote-522 trial combination of carboplatin/taxane-anthracycline NACT with the anti-PD1-antibody pembrolizumab (PEM) has been shown to be associated with a significantly higher pCR and clinically meaningful better EFS and a trend to better OS. Noteworthy only patients with more advanced stages IIa-III TNBC were included into the Keynote-522 trial. Although this effect was independent of clinically assessed nodal status, there is still some uncertainty on the optimal treatment in patients with clinical stage I.

In the metastatic setting, SG as a Trop-2-antibody-drug-conjugate has been shown to be highly efficacious in severely pre-treated patients (all with A/T pre-treated tumours, most of them carboplatin and 1/3 also anti-PD1 pre-treated) compared to chemotherapy of investigator´s choice. Treatment with SG was associated with significant longer median PFS (5.5 vs. 1.7 months) and longer median OS (12.1 vs. 6.7 months). Objective response was dramatically higher in the SG group vs. treatment by physician´s choice group (34.9 vs. 4.7%), in particular in the 2nd-3rd-line therapy (40% vs. 4%). Moreover, Tropics-02 trial has shown higher efficacy of SG vs. chemotherapy of investigator´s choice in patients with HR-positive/HER2-negative metastatic breast cancer.

In the neoadjuvant setting, recently presented results from the NeoSTAR trial show a promising pCR-rate of 30% and RCB 0-1-rate of 36% in TNBC patients with mostly stage II-III-disease (about 80%) after only 4 cycles of SG.

The following clinical questions are of highest medical need

1. Can 12-18 weeks neoadjuvant treatment with SG alone or in combination with PEM be associated with comparable pCR-rates (but more favourable safety profile) as shown for polychemotherapy in TNBC patients at lower relapse risk in historical controls?
2. Can SG-based therapy, as the most promising agent in patients with chemo-resistant disease, be associated with a such better prognosis (measured by 3-year-iDFS) compared to historical controls, which would make a randomized phase III-trial obsolete?

ELIGIBILITY:
Inclusion Criteria:

1. ER + PR negative or low positive (≤10% positive cells in IHC), and HER2 negative (i.e., IHC 0 - 1+ or IHC 2+ with FISH negative) breast cancer
2. All patients, independent from gender
3. ≥18 years at diagnosis
4. Histologically confirmed unilateral, primary invasive carcinoma of the breast Note: bilateral, multicentric, or multifocal carcinoma may be included, if there is a clear target lesion, that is subject to treatment decisions and solely evaluated and documented for study purposes.
5. Clinical stage I: cT1a-c, cN0 (clinical stage II only, if patient does not qualify for neoadjuvant polychemotherapy+PEM, e.g., elderly population, per investigator´s decision)
6. No clinical evidence for distant metastasis (M0)
7. Tumour block available for central pathology review
8. Performance Status ECOG ≤ 1 or KI ≥ 80%
9. Negative pregnancy test (urine or serum) within 7 days prior to registration in premenopausal patients
10. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
11. The patient must be willing and able to comply with the requirements and restrictions in this protocol and accessible for treatment and follow-up
12. Laboratory requirements:

    * Leucocytes ≥3.5 109/L,
    * Neutrophils > 1.5 109/L,
    * Platelets ≥100 109/L,
    * Haemoglobin ≥10 g/dL,
    * AP < 5.0 ULN,
    * AST ≤2.5 x ULN,
    * ALT ≤2.5 x ULN,
    * Total bilirubin ≤1 x ULN,
    * Creatinine ≤1.5 × ULN OR clearance ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
13. Clinical assessments:

    • LVEF within normal limits of each institution, measured by echocardiography and normal ECG (within 42 days prior to treatment)
14. The following age-specific requirements apply:

    * Women aged <50 years will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the site.
    * Women aged ≥ 50 years will be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments.
15. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods outlined for women of child-bearing potential if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to randomization/study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
16. Female patients of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception, presented in Table 1 (see Section 4.4.2), from the time of screening and must agree to continue using such precautions for 7 months after the last dose of IMP. Not all methods of contraception are highly effective. Female patients must refrain from breastfeeding while on study and for 7 months after the last dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic, or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable.
17. Female patients must not donate, or retrieve for their own use, ova from the time of randomisation and throughout the study treatment period, and for at least 7 months after the final study drug administration. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to enrolment in this study.
18. A male participant must agree to use a contraception as detailed in Appendix C of this protocol during the treatment period and for at least 7 months after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

1. Known hypersensitivity reaction to the compounds or incorporated substances of the IMPs
2. Prior malignancy with a disease-free survival of < 5 years, except curatively treated basalioma of the skin or pTis of the cervix uteri
3. Any history of invasive breast cancer
4. Previous or concurrent treatment with cytotoxic agents for any non-oncological reason unless clarified with sponsor
5. Concurrent treatment with other experimental drugs
6. Participation in another interventional clinical trial with or without any investigational not marketed drug within 30 days prior to study entry
7. Concurrent pregnancy; patients of childbearing potential or potentially childbearing partners of male patients must implement a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
8. Breast feeding woman
9. Reasons indicating risk of poor compliance
10. Patients not able to consent
11. Known polyneuropathy ≥ grade 2
12. Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study including recovery from major surgery, autoimmune disease, known psychiatric/substance abuse disorders, acute cystitis, ischuria, and chronic kidney disease
13. Uncontrolled infection requiring i.v. antibiotics, antivirals, or antifungals
14. History of pneumonitis
15. Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients should be tested for HIV prior to randomisation if required by local regulations or ethics committee (EC).
16. Have active hepatitis B virus (HBV) or hepatitis C virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.

    * Patients who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
    * Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require a HCV antibody at screening and will only require HCV RNA by quantitative PCR for confirmation of active disease.
17. Patients who test positive for HIV antibody.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
pathological complete remission (pCR) | at surgery
  no invasive tumour in breast and lymph nodes (ypT0/is and ypN0)
invasive disease-free survival rate (iDFS), | after 3 years
  time from date of first diagnosis to any invasive breast cancer event, death or secondary malignancy according to STEEP 2.0 criteria

SECONDARY OUTCOMES:
Overall survival (OS) | 6 years
  time from first diagnosis to death
distant disease-free survival (dDFS) | after 3 years
  distant disease-free survival
distant disease-free interval (dDFI) | after 3 years
  distant disease-free interval
recurrence-free survival (RFS) | after 3 years
  recurrence-free survival
local recurrence-free survival (LRFS) | after 3 years
  local recurrence-free survival
Breast cancer free interval (BCFI) | after 3 years
  Breast cancer free interval
Health-related Quality of Life: Quality of Life Questionnaire C30 | Baseline to end of cycle 2 (each cycle is 21 days)
  change in QLQ-C30-Score; min 0 - max 100 points; the higher the better quality of life
Health-related Quality of Life: Quality of Life Questionnaire BR45 | Baseline to end of cycle 2 (each cycle is 21 days)
  change in BR45-Score; min 0 - max 100 points; the higher points on functional scale the better the function; the higher points on symptom scale the higher the symptomatology.
Health-related Quality of Life: Quality of Life Questionnaire C30 | Baseline to end of cycle 4 (each cycle is 21 days)
  change in QLQ-C30-Score; min 0 - max 100 points; the higher the better quality of life
Health-related Quality of Life: Quality of Life Questionnaire BR45 | Baseline to end of cycle 4 (each cycle is 21 days)
  change in BR45-Score; min 0 - max 100 points; the higher points on functional scale the better the function; the higher points on symptom scale the higher the symptomatology.
Health-related QoL: EORTC QLQ-C30 | Baseline to end of cycle 6 (each cycle is 21 days)
  change in QLQ-C30-Score; min 0 - max 100 points; the higher the better quality of life
Health-related Quality of Life: Quality of Life Questionnaire BR45 | Baseline to end of cycle 6 (each cycle is 21 days)
  change in BR45-Score; min 0 - max 100 points; the higher points on functional scale the better the function; the higher points on symptom scale the higher the symptomatology.
Health-related QoL: EORTC QLQ-C30 | Baseline to timepoint before surgery
  change in QLQ-C30-Score; min 0 - max 100 points; the higher the better quality of life
Health-related QoL: EORTC QLQ-BR45 | Baseline to timepoint before surgery
  change in QLQ-BR45-Score
Health-related Quality of Life: Quality of Life Questionnaire C30 | Baseline to timepoint 1 year after surgery
  change in QLQ-C30-Score; min 0 - max 100 points; the higher the better quality of life
Health-related Quality of Life: Quality of Life Questionnaire BR45 | Baseline to timepoint 1 year after surgery
  change in BR45-Score; min 0 - max 100 points; the higher points on functional scale the better the function; the higher points on symptom scale the higher the symptomatology.

OTHER OUTCOMES:
Other pCR-definitions | at time of surgery
  ypT0/is, any ypN
  * ypT0, ypN0
  * near pCR (ypT1a/is, any ypN)
stromal tumour infiltrating lymphocytes (sTIL) | at baseline and after 3 weeks of therapy
  percentage of sTIL

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, Prof Dr PHD, Principal Investigator — Westdeutsche Studiengruppe GmbH; Nadia Harbeck, Prof Dr, Principal Investigator — Breast Centre, Dept. Obstetrics & Gynaecology and CCC Munich LMU University Hospital; Oleg Gluz, PD Dr, Principal Investigator — Breast Centre, Evang. Bethesda-Hospital, Moenchengladbach; Sherko Kuemmel, Prof Dr, Principal Investigator — Breast Centre, Kliniken Essen Mitte; Monika Graeser, PD Dr.., Principal Investigator — Breast Centre, Evang. Bethesda-Hospital, Moenchengladbach
Locations (42):
- Germany (42):
  - Stadtklinik Baden-Baden / Brustzentrum, Baden-Baden, Baden-Wurttemberg
  - Kliniken Böblingen, Böblingen, Baden-Wurttemberg
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau, Baden-Wurttemberg
  - SLK Kliniken Heilbronn, Frauenklinik, Heilbronn, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - GRN Klinik Weinheim, Weinheim, Baden-Württembergs
  - Hämatologie-Onkologie im Zentrum MVZ GmbH, Augsburg, Bavaria
  - Universitätsklinikum Augsburg A.ö.R., Augsburg, Bavaria
  - Rotkreuzklinikum München, München, Bavaria
  - DBZ Onkologie GmbH, Berlin, Brandenburg
  - Klinikum Ernst von Bergmann gGmbH, Potsdam, Brandenburg
  - Klinikum Bremerhaven Reinkenheide gGmbH, Bremerhaven, City state Bremen
  - AGAPLESION Markus Krankenhaus, Frankfurt am Main, Hesse
  - MVZ II der Niels Stensen Kliniken, Georgsmarienhütte, Lower Saxony
  - Gynäkologische Gemeinschaftspraxis-Ärztehaus am Bahnhofsplatz, Hildesheim, Lower Saxony
  - Ev. Krankenhaus Berlin-Spandau, Berlin, North Rhine-Westphalia
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld, North Rhine-Westphalia
  - St. Elisabeth-Krankenhaus Köln-Hohenlind, Cologne, North Rhine-Westphalia
  - Kliniken der Stadt Köln, Krankenhaus Holweide, Cologne, North Rhine-Westphalia
  - MVZ Medical Center Düsseldorf - GynOnco, Düsseldorf, North Rhine-Westphalia
  - St. - Antonius - Hospital, Eschweiler, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - ev. Klinikum Gelsenkirchen - Klinik für Senelogie, Gelsenkirchen, North Rhine-Westphalia
  - St. Barbara Klinik Hamm GmbH, Hamm, North Rhine-Westphalia
  - Klinikum Leverkusen gGmbH, Leverkusen, North Rhine-Westphalia
  - Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, North Rhine-Westphalia
  - MVZ MediaVita, St. Franziskus-Hospital Münster, Münster, North Rhine-Westphalia
  - MKS St.Paulus GmbH (ehem.Marienkrankenhaus), Schwerte, North Rhine-Westphalia
  - Praxisnetzwerk Hämatologie und Onkologie, Troisdorf, Troisdorf, North Rhine-Westphalia
  - Marien Hospital Witten, Witten, North Rhine-Westphalia
  - Helios Universitätsklinikum Wuppertal Barmen, Wuppertal, North Rhine-Westphalia
  - Klinikum Mutterhaus-Trier, Trier, Rhineland-Palatinate
  - Caritasklinikum Saarbrücken, Saarbrücken, Saarland
  - Johanniter GmbH Johanniter Krankenhaus Stendal, Stendal, Sachsen-Anhalts
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Charité Campus Mitte Universitätsklinikum Berlin, Berlin
  - Hämatologisch/Onkologische Schwerpunktpraxis Bremen, Bremen
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
  - Klinikum der Universität München, München

IPD SHARING:
Plan to Share IPD: No